CLINICAL TRIAL: NCT01521299
Title: A Phase I Dose Escalation Study of Hydroxyurea in Combination With SCH900776 in Advanced Malignant Solid Tumors
Brief Title: A Dose Escalation Study of Hydroxyurea in Combination With SCH900776 in Advanced Malignant Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient population of eligible patients.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1049
Record Dates: First submitted 2011-10-31; First posted 2012-01-30 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Advanced Solid Tumors
Keywords: hydroxyurea; S phase; G2 phase; pharmacokinetics
MeSH Terms: interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hydroxyurea — oral hydroxyurea on days 1,8 and 15

SUMMARY:
This is an open label Phase I study with two parts. Part Two with SCH900776 in combination with hydroxyurea will not be pursued at this time.

Part One investigates monotherapy with oral hydroxyurea. The primary objective is to determine whether a tolerated dose (TD) of hydroxyurea as a single agent can increase the percentage of tumor cells in S and G2 phase of the cell cycle. For this reason, all patients in Part One must have a tumor lesion accessible for a skin punch biopsy. Tumor biopsies will be obtained on two separate occasions: prior to hydroxyurea and at 16-18h after starting hydroxurea therapy on day 1 only.

A baseline 12-lead ECG will be obtained from each study participant. Single-agent hydroxyurea will be administered on days 1, 8 and 15 of a 28 day cycle, for ONE cycle only. On these days oral hydroxyurea will be started in the late afternoon and administered every 4 hours for a total of 6 doses.

Venous (up to 10 mL) blood samples will be obtained at time zero (pretreatment), 30 min, 1h, 1.5 2, 2.5, 3.0, 3.5 and 4h following the first oral dose of hydroxyurea, and pretreatment and at the same times following the sixth oral dose of hydroxyurea (i.e., 20, 20.5, 21, 21.5, 22, 22.5, 23, 23.5 and 24 h).

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or metastatic, histologically/cytologically confirmed malignant solid tumors or lymphoma which has progressed on standard therapy.
2. Study participants must have a Karnofsky Performance status of > 70.
3. Study participants must have a predicted life expectancy of at least 3 months.
4. Study participants must have measurable or evaluable disease.
5. Study participants must be at least 18 years.
6. Study participants (and/or parent/guardian for study participants who are otherwise unable to provide independent consent) must be willing and able to give written informed consent and adhere to study visit schedules.
7. A female study participant of child-bearing potential or a male study participant and their female sexual partner(s) of child-bearing potential who are sexually active must agree to use a medically accepted method of contraception prior to enrollment while receiving protocol-specified medication and for 6 months after stopping the medication. Acceptable methods of contraception include double-barrier methods such as male or female condom in combination with spermicides, or diaphragm or cervical cap with spermicides, or medically prescribed intrauterine device. Contraceptive medication (i.e. oral contraceptives) vasectomy and tubal ligation should each be considered a single barrier.
8. A female study participant of child-bearing potential or a male subject and their female sexual partner(s) of child-bearing potential who are not currently sexually active must agree to use a medically accepted method of contraception should they become active while participating in the study.
9. Premenopausal women will require a negative pregnancy test within 7 days of study entry.
10. Study participants must have adequate renal function as evidenced by an estimated creatinine clearance (eCrCl using the Cockcroft-Gault formula) of > 60 mL/min.
11. Study participants must have adequate bone marrow function as evidenced by absolute neutrophil counts (ANC) ≥ 1500 µL, and platelet counts ≥100,000 µL.
12. Study participants, except those with Gilbert's Syndrome, must have adequate hepatic function as evidenced by serum total bilirubin ≤ 1.5 x ULN and AST/ALT levels ≤ 2.5 x ULN for the reference laboratory. If the study participant has known hepatic metastatic disease then AST/ALT should be ≤ 5.0 x ULN.
13. Tumor site accessible for both pre-treatment and post-treatment biopsies will be required for a minimum of 67% of study participants in each dose cohort where "n" is at least 3. In PART ONE of the study the first cohort-dose level 0, (who will receive hydroxyurea plus zero mg of SCH900776) is unique in that all participants in this cohort will be required to have biopsiable tumor sites.

EXCLUSION CRITERIA:

1. Study participant has a known hypersensitivity to hydroxyurea or SCH900776 or to any of their excipients/diluents.
2. Study participant has received any medication listed in Section 4.3 more recently than the indicated washout period prior to the receiving the first dose of SCH900776
3. Study participant has known history of or behavior predisposing to human immunodeficiency virus (HIV) infection, active hepatitis B or hepatitis C, or liver cirrhosis or active ethanol abuse
4. Study participant is New York Heart Association (NYHA) Class III (has marked limitation in activity due to symptoms, even during less-than-ordinary activity [i.e. walking short distances > 20 to 100 m]; or being comfortable only at rest) or Class IV (has severe limitations; experiences symptoms even while at rest; mostly bed bound)
5. Study participant has any other medical or psychiatric condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial
6. Study participant has undergone major surgery within 3 weeks prior to first study drug treatment
7. Study participant has central nervous system (CNS) or leptomeningeal metastases
8. Study participant has any of the following within 6 months prior to starting the first study drug treatment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or seizure disorder
9. Study participant has known congenital or acquired bleeding diathesis, e.g. hemophilia.
10. Study participant has baseline QTcB > 480 msec women, QTcB > 470 msec men (i.e. CTACAE v 4.0 Grade ≥ 2) (This exclusion criteria may be removed/modified based on SCH900776 Phase I safety and evolving QTc study findings)
11. Study participant is currently a heavy smoker and/or is likely to continue heavy smoking during the study (a heavy smoker is defined as smoking > 10 cigarettes/day)
12. Female study participant is breast feeding, pregnant or intends to become pregnant
13. Study participant is participating in any other cancer chemotherapy treatment clinical study
14. Study participant participation in another non-interventional study may be considered after discussion between the Principal Investigator and the SCH900776 IND holders Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of tumor cells in S and G2 phase of the cell cycle | 16 hours post dose.
  A tissue biopsy is collected at 16 hours post dose.

SECONDARY OUTCOMES:
Blood concentrations of single agent hydroxyurea at multiple timepoints. | Blood samples are collected within 24 hours of initial hydoroxyurea dose.
  Pharmacokinetic-pharmacodynamic modeling of drug concentrations/exposure to tumor molecular pharmacodynamics will be done using appropriate Emax or sigmoid Emax direct PK-PD models. Blood samples: time 0 (pretreatment), 30 min, 1h, 1.5 2, 2.5, 3.0, 3.5 and 4h following the first oral dose of hydroxyurea, and pretreatment and at the same times following dose 6 (i.e., 20, 20.5, 21, 21.5, 22, 22.5, 23, 23.5 and 24 h)

CONTACTS AND LOCATIONS:
Overall Officials: Margit M McGowan, DO, Principal Investigator — Dartmouth-Hitchcock Medical Center